CLINICAL TRIAL: NCT00696722
Title: Influence of Atazanavir Treatment on Endothelial Dysfunction, Vascular Inflammation and Heme Oxygenase Activity in Type 2 Diabetes Mellitus
Brief Title: Effects of Atazanavir Treatment on Type 2 Diabetes Mellitus Related Endothelial Dysfunction
Acronym: DM2ATV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Diabetes Research Foundation (Other)
Responsible Party: P. Smits, Radboud University Nijmegen Medical Centre
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DM2ATV; 2006.00.055
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2009-01

CONDITIONS: Type 2 Diabetes Mellitus Related Endothelial Dysfunction
MeSH Terms: interventions — Atazanavir Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): Placebo treatment first, atazanavir treatment second
  Interventions: Drug: placebo + atazanavir
- 2 (Experimental): Atazanavir treatment first, placebo treatment second
  Interventions: Drug: atazanavir + placebo

INTERVENTIONS:
Drug: placebo + atazanavir — Placebo treatment first, atazanavir treatment second
  4 day treatment
  Arms: 1
Drug: atazanavir + placebo — Atazanavir treatment first, placebo treatment second
  4 day treatment
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether atazanavir use is of influence on the endothelial dysfunction associated with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria (most important):

* 18 - 70 years
* type 2 diabetes mellitus treated with diet, oral medication and/or insulin
* BMI of 18 to 35
* determinants of renal and hepatic function within twice the upper limit of normal range, abnormalities in lipid profile permitted

Exclusion Criteria (most important):

* history of smoking within past year
* history of or current abuse of drugs, alcohol or solvents
* current use of antihypertensive, cardiac or other vasoactive medication
* clinical evidence of cardiac or pulmonary disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Acetylcholine induced vasodilation | following a 4 day treatment with either placebo or atazanavir

SECONDARY OUTCOMES:
heme oxygenase expression and activity | following a 4 day treatment with either placebo or atazanavir
assessment of vascular inflammation by determination of adhesion molecule levels | following a 4 day treatment with either placebo or atazanavir

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands